CLINICAL TRIAL: NCT05712499
Title: Investigation of the Effect of Mindfulness-based Psychoeducation on Defense Mechanisms and Mindful Awareness in Nursing Students
Brief Title: Mindfulness-based Psychoeducation and Defense Mechanisms, Mindful Awareness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Burcu Demir Gokmen, Associate Professor, Agri Ibrahim Cecen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AICU-SBF-HB-BDG-01
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Mindfulness; Psychoeducation; Defense Mechanisms; Awareness

STUDY DESIGN:
Intervention Model Description: This study was designed as a quasi-experimental study with a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based psychoeducation program (Experimental): The group in which the mindfulness-based psychoeducation program was applied.
  Interventions: Behavioral: mindfulness-based psychoeducation program
- control group (Active Comparator): The group in which no intervention was made and only the pre-test and post-test were applied for comparison.
  Interventions: Behavioral: ongoing life

INTERVENTIONS:
Behavioral: mindfulness-based psychoeducation program — Mindful awareness is a mind and body practice that involves increasing attention to what is happening at the moment and accepting what is perceived without judgment. Mindfulness includes awareness and attention; Awareness is the mechanism that constantly controls the of the state of consciousness. Mindfulness-based cognitive therapies are evidence-based psychoeducation. Psychoeducation was organized in 2 consecutive sessions once a week for 8 weeks, and each session was 60 minutes, in total 16 sessions. The content of the psychoeducation program was explained in detail, and techniques such as presentation and question-answer narrative techniques, video, audio recording, mindfulness assignments for the next session were used in the training.
  Arms: Mindfulness-based psychoeducation program
Behavioral: ongoing life — The control group continued with their lives without any intervention. Only pre-test and post-test were applied. While the program was applied to the experimental group, no intervention was made to the control group.
  Arms: control group

SUMMARY:
Purpose: Nowadays, it is seen that there is an increasing interest in mindfulness-based therapies. Such practices can be beneficial by contributing to the personal and professional development of nursing students. In the study, the effect of mindfulness-based psychoeducation applied to Turkish nursing students on defense mechanisms and mindfulness was evaluated.

Method: The research was designed as a quasi-experimental study with a control group. The population of the study consisted of 96 newly enrolled students in the nursing department of a foundation university, and the sample consisted of a total of 72 students who met the inclusion criteria of the study. In the sample, while 33 students formed the intervention group, 39 students formed the control group. Mindfulness- Based Psychoeducation was given online in 16 sessions in 8 weeks. Data were collected using the Defense Style Questionnaire and the Awareness Scale.Percentage distributions were used in the analysis of the data, t-Test and Chi-Square test were used in the comparison of the intervention and control groups, and the paired-samples t-Test was used in the comparison of the intervention and control groups within the group.

DETAILED DESCRIPTION:
Population-Sample It was conducted with 96 nursing students enrolled in the Faculty of Health Sciences of a state university in the east of Turkey in the 2020-2021 academic year. 86 students who met the research criteria (being a first-year student, being over the age of 18, not having any psychiatric diagnosis, volunteering to participate in the study, not having received mindfulness training before, not a foreign national) were included in the study. It was deemed appropriate to participate in the study by first-year students who were at the beginning of their nursing education and had not yet taken a course related to personal development (such as introduction to psychology, interpersonal relations and communication). Among these students, the intervention and control groups were formed after detailed information about the research process was given according to students' requests, without being randomized. Those who wanted to receive training and believed that they could attend the training continuously were determined as the intervention group (45), and those who did not want to participate in the training and were unsure were determined as the control group (41). However, the research was completed with 33 students in the intervention group and 39 students in the control group. 12 students from the intervention group left the research because they could not attend the sessions regularly, while 2 students in the control group left the research without stating a reason for their request. In the power analysis of 72 students participating in the research.

Data Collection and Program Application Due to the Covid-19 pandemic, nursing education was continued in our institution in the 2020-2021 academic year with a distance education called DEP(Distance Education Platform). This situation necessitated online psychoeducation to be given as part of the research. The Mindfulness-Based Psychoeducation program was conducted via DEP(Distance Education Platform)between 08.03.2021 and 30.04.2021 after obtaining the necessary permission and support from the institution. The scales created by the researcher through "Google Form" were shared with the students in the Mindfulness-Based Psychoeducation Program at DEP(Distance Education Platform)and the pretest data were collected in the first session, whereas the posttest data were collected two weeks after the last session. On the first page of this form, the purpose of the research was explained, the confirmation icon indicating that they voluntarily accepted to participate in the research, why they had to give name or code information, and the response time (30 minutes) for the forms were stated.

Data Collection Tools This study, Personal Information Form, Defense Style Questionnaire (DSQ-40), and Mindful Attention Awareness Scale (MAAS) were used.

Personal Information Form It consists of questions about the sociodemographic characteristics of the students (age, gender).

Defense Style Questionnaire (DSQ-40) In the scale, which determines the appearance of defense mechanisms at the level of consciousness and behavior, and consists of 40 items, 20 defenses, and 3 sub-dimensions (mature, neurotic, and immature), each item is evaluated between 1-9 (absolutely inappropriate - absolutely appropriate). Mature defenses are; suppression, anticipation, sublimation, and humor. Neurotic defenses; subversion, counter-reaction, idealization, and artificial altruism. Immature defenses are; passive aggression, expression, projection, isolation, denial, division, devaluation, autistic fantasy, displacement, dissociation, rationalization, and somatization. The scale is scored on defenses or sub-dimensions, not on the total score. Total score or arithmetic mean is used while calculating each defense or sub-dimension. As the score increases, the use of the defense/sub-dimension also increases. In the Turkish adaptation study of the scale, the Cronbach's Alpha values were 0.70, 0.61, and 0.83, respectively, according to the mature, neurotic, and immature sub-dimensions whereas in this study, it was 0.65, 0.71, and 0.82.

Mindful Attention Awareness Scale (MAAS) The scale has a 15-item and 6-point Likert feature that measures the differences in the ability to be aware of what is happening in the moment and to pay attention to them. The scores obtained from the scale vary between 15-90 points. A high score indicates a high level of mindful awareness. While the Cronbach Alpha value of the scale was 0.80 in the Turkish adaptation study, it was 0.82 in this study.

Mindfulness-based psychoeducation program Mindfulness-based cognitive therapies are evidence-based psychoeducation. Psychoeducation was organized in 2 consecutive sessions once a week for 8 weeks, and each session was 60 minutes, in total 16 sessions. The content of the psychoeducation program was explained in detail, and techniques such as presentation and question-answer narrative techniques, video, audio recording, mindfulness assignments for the next session were used in the training. A Whatsapp group was created to remind and share materials with students participating in psychoeducation. It was stated that the students should be very careful, observant, and patient while doing the practices to get to know themselves, be aware of their emotions, thoughts, bodily sensations and focus. The applications were performed online-live in DEP(Distance Education Platform)and recorded by the system. The researcher's camera was turned on and the students' camera was also left to preference. The privacy of all participants was given importance and it was stated that the existing recordings would not be used anywhere else, that the participants would not be able to take recordings, and that the sharing in the sessions should be kept confidential. The students were able to access the records at any time during the day that the psychoeducation started and for 15 days after the end of the psychoeducation. In the days when there is no psychoeducation, reminder messages were sent twice a week via and DEP(Distance Education Platform) applications for home applications.

Evaluation of Data The coding and analysis of the data were done via the SPSS-23( Statistical Package for the Social Sciences-23) program, and the significance level was accepted as p<0.05. Percentage distributions were used in the analysis of the data, t-Test and Chi-Square test were used in the comparison of the intervention and control groups, and the paired-samples t-Test was used in the comparison of the intervention and control groups within the group.

Declarations The necessary institutional permission and support for the research were obtained from the Deanery of the Faculty of Health Sciences. In addition, ethical permission was obtained from the Ethics Committee of the Institute of Health Sciences of the University. (Decision dated 27.01.2021 and numbered 2021/18). Oral and written informed consent was obtained from the students participating in the research and the research was conducted following the Principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Without a psychiatric diagnosis,

  * Have not done awareness practices before,
  * Not meditating,
  * Not a foreign national,
  * Those who volunteered to participate in the study

Exclusion Criteria:

-

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Change of defense mechanisms level after 10 weeks. | baseline and 10 weeks.
  Defense Style Questionnaire (DSQ-40) : In the scale, which determines the appearance of defense mechanisms at the level of consciousness and behavior, and consists of 40 items, 20 defenses, and 3 sub-dimensions (mature, neurotic, and immature), each item is evaluated between 1-9 (absolutely inappropriate - absolutely appropriate)The scale is scored on defenses or sub-dimensions, not on the total score. Total score or arithmetic mean is used while calculating each defense or sub-dimension. As the score increases, the use of the defense/sub-dimension also increases.
Change of mindful awareness level after 4 weeks. | baseline and 10 weeks.
  Mindful Attention Awareness Scale (MAAS):The scale has a 15-item and 6-point Likert feature that measures the differences in the ability to be aware of what is happening in the moment and to pay attention to them. The scores obtained from the scale vary between 15-90 points. A high score indicates a high level of mindful awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Demir Gokmen, phd, Principal Investigator — Agri Ibrahim Cecen Universty
Locations (1):
- Agri Ibrahim Cecen Universty /Faculty of Health Sciences, Ağrı, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is a plant for the use of other customers in the individual loading body (IPD).